CLINICAL TRIAL: NCT03963947
Title: Observational Prospective Study to Assess the Safety and Effectiveness of Beltavac® Polymerized With House Dust Mites
Brief Title: Study to Assess the Safety and Effectiveness of Beltavac® Polymerized With House Dust Mites
Status: Completed | Type: Observational
Sponsor: Alfons Malet i Casajuana (Other)
Collaborators: Probelte Pharma S.L.U. (Industry)
Responsible Party: Sponsor-Investigator, Alfons Malet i Casajuana, Head of Allergy Service in Teknon Medical Center, Centro Medico Teknon
Organization: Centro Medico Teknon (Other)
Other Study IDs: MAL-BEL-2018-01
Record Dates: First submitted 2019-05-23; First posted 2019-05-28 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Rhinoconjunctivitis With or Without Allergic Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Beltavac® Polymerized with house dust mites — Adminstration of Beltavac® Polymerized with house dust mites according to the routine clinical practice

SUMMARY:
Non-interventional Study to Assess the Safety and Effectiveness Profile of a SCIT Therapy With Beltavac® Polymerised With House Dust Mite in pediatric allergic patients

DETAILED DESCRIPTION:
This prospective open multi-center non-interventional study assess the safety and effectiveness profile of the subcutaneous allergen-specific immunotherapy with Beltavac polymerized with house dust mite pediatric allergic patients in routine medical care.

Patients receive a rush schedule administration every month for a year. They attend at least 5 study visits to inform about the adverse reactions, the self reported symptoms and the medication intake.

ELIGIBILITY:
Inclusion Criteria:

* Patients from 3 to 11 years suffering from a clinically relevant Dermatophagoides farinae and Dermatophagoides pteronyssinus induced allergic rhinitis or rhinoconjunctivitis associated with or not with asthma
* Positive skin testing
* Positive Serum-Specific IgE determination
* Parental or legal representative informed consent
* Clinical sintomatology on the inclusion period

Exclusion Criteria:

* Patients suffering from acute or chronic infections or inflammations
* Patients suffering from uncontrolled and severe asthma
* Patients with a known autoimmune disease
* Patients with active malignant disease
* Patients requiring beta-blockers
* Patients having any contraindication for the use of adrenaline
* Patients with previous immunotherapy with this allergen or another allergen with cross-reaction
* Patients with immunotherapy treatment at the time of inclusion

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients from 3 to 11 years, who suffer from allergic rhinitis or rhinoconjunctivitis associated with or not with asthma caused by house dust mites
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2023-05-24 (Actual); Study Completion 2023-05-24 (Actual)

PRIMARY OUTCOMES:
Numbers of treatment-related local and systemic reactions | 1 Year

SECONDARY OUTCOMES:
Combined symtom and medication score of Rhinoconjunctivitis | 1 Year
  The score will be calculated as a sum of the symptoms score (0-3) and medication score (0-3)
Combined symtom and medication score of Asthma | 1 Year
  The score will be calculated as a sum of the symptoms score (0-3) and medication score (0-3)
Visual analogue Scale Score | 1 Year
  Psycometric scale that assesses the global allergic disease discomfort. It is a 10 cm line representing severity from 0:"no symptoms" to 10 "highest level of symptoms"
IgE and IgG4 specific quantification | 1 Year

CONTACTS AND LOCATIONS:
Locations (1):
- Teknon Medical Center, Barcelona, Spain